CLINICAL TRIAL: NCT00686478
Title: A Double-blind Placebo Controlled Trial Using Subcutaneous Injections of Intron A for the Treatment of Hypertrophic Scar
Brief Title: Intron A for the Treatment of Hypertrophic Scar
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial is not being done at this time
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Ted Tredget, Principal Investigator, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IFN - 1598
Record Dates: First submitted 2008-05-26; First posted 2008-05-29 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Burn; Hypertrophic Scar
Keywords: burn; hypertrophic scar; fibroproliferative disorder
MeSH Terms: conditions — Burns; Cicatrix, Hypertrophic | interventions — Interferon alpha-2; Introns

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- interferon alpha 2b (Intron A) (Experimental): 1 million IU of interferon alpha 2b (Intron A) subcutaneously once a day for 7 days, then 3 million IU of interferon alpha 2b (Intron A) subcutaneously three times a week for 23 weeks.
  Interventions: Drug: interferon alpha 2b
- Placebo (Placebo Comparator): Placebo administered subcutaneously once a day for 7 days, then three times a week for 23 weeks.
  Interventions: Drug: interferon alpha 2b

INTERVENTIONS:
Drug: interferon alpha 2b — 1 million IU of interferon alpha 2b (Intron A) subcutaneously once a day for 7 days, then 3 million IU of interferon alpha 2b (Intron A) subcutaneously three times a week for 23 weeks.
  Other Names: intron a

SUMMARY:
This study assesses the intervention with antifibrotic agents, specifically interferon (IFN) to reduce the magnitude and duration of hypertrophic scar. Burn patients with hypertrophic scar are randomly assigned to either an intervention IFN group or a placebo control group by subcutaneous injection three times a week. Patients are assessed using cutometer, mexameter, standardized photography, urinalysis, blood work, tissue biopsies and the Vancouver Burn Scar Assessment (VBSA) which rates selected HTS based on color, vascularity, height, pliability, itchiness and pain sensitivity. Once on treatment patients are assessed monthly for the six month treatment period.

DETAILED DESCRIPTION:
Burn patients being followed and treated in the Outpatient Burn Clinic with large areas of HTS are approached to participate in the study. Patients who agree to participate and who have signed an informed consent are entered into the trial.

Pre-treatment evaluation and monthly examinations include:

* standardized photographs of scar
* scar volume
* Vancouver Burn Scar Assessment (VBSA)
* blood work (TGF-beta, histamine)
* urine collection (histamine)
* 6mm punch biopsy of HTS and adjacent normal skin (every two months)

Patients are randomized to received with placebo or Intron A 1x106 IU a day for 7 days, then 3x106 IU 3 SC, three times a week for 23 weeks.

ELIGIBILITY:
Inclusion Criteria:

* burns > 5% tbsa
* informed consent
* no prior exposure to interferon or other cytokines

Exclusion Criteria:

* history of cardiac or CNS disorder or disease
* autoimmune disease
* immunodeficiency
* abnormal renal or hepatic function
* pregnancy
* serious intercurrent illness
* active infection
* malnutrition
* active drug or alcohol abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Systemic effect of Intron A on hypertrophic scar | once / month for 6 months
  standardized photographs of scar, scar volume, Vancouver Burn Scar Assessment (VBSA), blood work (TGF-beta, histamine), urine collection (histamine), biopsy of HTS and adjacent normal skin.

CONTACTS AND LOCATIONS:
Overall Officials: Edward E Tredget, MD MSc FRCSC, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada